CLINICAL TRIAL: NCT00000255
Title: Differential Acute Tolerance Development to Effects of Nitrous Oxide
Brief Title: Differential Acute Tolerance Development to Effects of Nitrous Oxide - 7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08391-7; R01DA008391 (NIH); R01-08391-7
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; acute tolerance; subjective effects; analgesia; psychomotor; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Agnosia | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 0% Nitrous oxide (Placebo Comparator)
  Interventions: Drug: Nitrous oxide
- 10% nitrous oxide (Active Comparator)
  Interventions: Drug: Nitrous oxide
- 20% nitrous oxide (Active Comparator)
  Interventions: Drug: Nitrous oxide
- 30% nitrous oxide (Active Comparator)
  Interventions: Drug: Nitrous oxide
- 40% nitrous oxide (Active Comparator)
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To examine differential acute tolerance development to effects of nitrous oxide in humans.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1995-04; Primary Completion 1996-05 (Actual); Study Completion 1996-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity, pain bothersomeness | 25, 70, & 115 min of inhalation and 40 min post
  Subjects will inhale varying conc of nitrous oxide for 120 min with cold immersion of forearm at 25, 70, and 115 min and 40 min after inhalation. Pain intensity and bothersomeness will be assessed at each immersion.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Zacny JP, Cho AM, Coalson DW, Rupani G, Young CJ, Klafta JM, Klock PA, Apfelbaum JL. Differential acute tolerance development to effects of nitrous oxide in humans. Neurosci Lett. 1996 May 10;209(2):73-6. doi: 10.1016/0304-3940(96)12626-4. PMID 8761985